CLINICAL TRIAL: NCT01291914
Title: A Double-Blind, Randomized,Placebo-Controlled, Two-Phase Study (a Single Ascending Dose Phase Followed by a Proof of Concept Phase) to Assess the Safety, Efficacy and Pharmacokinetics of FX005 for the Treatment of Pain in Osteoarthritis of the Knee
Brief Title: Study of FX005 for the Treatment of Pain in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX005-2010-001
Record Dates: First submitted 2011-02-04; First posted 2011-02-09 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; knee; intra-articular; safety; efficacy; pharmacokinetics; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Carrier State

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FX005 (Experimental)
  Interventions: Drug: FX005
- Placebo 1 (Carrier) (Placebo Comparator)
  Interventions: Drug: Placebo 1 (Carrier)
- Placebo 2 (Diluent) (Placebo Comparator)
  Interventions: Drug: Placebo 2 (Diluent)

INTERVENTIONS:
Drug: FX005 — Single Ascending Dose (SAD) Phase Cohorts: 1, 10 or 45 mg intra-articular injection; Proof of Concept Phase: Maximum, well-tolerated dose intra-articular injection (determined during SAD Phase)
  Arms: FX005
Drug: Placebo 1 (Carrier) — Single intra-articular injection
  Arms: Placebo 1 (Carrier)
Drug: Placebo 2 (Diluent) — Single intra-articular injection
  Arms: Placebo 2 (Diluent)

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy and pharmacokinetics of FX005 for the treatment of pain in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
The objectives of the study are to assess FX005, as compared to placebo control, for:

* Safety and tolerability
* Analgesic effect
* Pharmacokinetics

Analgesic effect will be assessed using the Western Ontario & McMaster University Osteoarthritis Index (WOMAC), the Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP) questionnaire, and patient and clinical observer global assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥40 years of age
* Diagnosis of unilateral or bilateral osteoarthritis of the knee for at least 6 months; confirmation of osteoarthritis according to American College of Rheumatology Criteria (clinical and radiological)
* Kellgren-Lawrence grades II or III
* Mean score for the WOMAC A subscale (pain) between 2.0 and 3.5 for the index knee
* Score of 2-3 for the WOMAC A1 score (pain on walking) for the index knee
* Body mass index ≤ 40 kg/m2
* Willingness to abstain from use of restricted medications during the study
* Willingness and ability to comply with the study procedures and visit schedule

Exclusion Criteria:

* Kellgren-Lawrence Grade 0, I or IV radiographic stage of the index knee
* Clinically apparent tense effusion in index knee
* Presence of surgical hardware or other foreign body in the index knee
* Clinical signs and symptoms of active knee infection or crystal disease
* Intra-articular corticosteroid within 3 months of Screening
* Intra-articular hyaluronic acid within 6 months of Screening
* Other intra-articular therapy within 3 months of Screening
* Prior arthroscopic or open surgery of the index knee within 12 months of Screening
* Planned/anticipated surgery of the index knee during the study period
* History of malignancy or other serious, non-malignant, significant, acute or chronic medical (e.g.. uncontrolled diabetes) or active psychiatric illness
* Skin breakdown at the knee where the injection would take place
* Women who are pregnant, nursing or likely to become pregnant during the time of the study
* Women of child-bearing potential (not surgically sterile or post-menopausal for at least 1 year) not using effective contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-12; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the WOMAC A score (pain subscale) | at 4 weeks post treatment

SECONDARY OUTCOMES:
Change from baseline in WOMAC A score (pain subscale) | over 4, 8 and 12 weeks post treatment
Change from baseline for WOMAC A score (pain subscale) | at 2, 8 and 12 weeks post treatment
Change from baseline for WOMAC B score (stiffness subscale) | at 2, 4, 8 and 12 weeks post treatment
Change from baseline for WOMAC C score (function subscale) | at 2, 4, 8 and 12 weeks post treatment
Change from baseline for WOMAC A1 response (pain on walking) | at 2, 4, 8 and 12 weeks post treatment
Change from baseline for WOMAC A1 response (pain on walking) | over 4, 8 and 12 weeks post treatment
Change from baseline for WOMAC total score | at 2, 4, 8 and 12 weeks post treatment
Change from baseline for ICOAP intermittent pain score | at 2, 4, 8 and 12 weeks post treatment
Change from baseline for ICOAP constant pain score | at 2, 4, 8 and 12 weeks post treatment
Change from baseline for ICOAP total score | at 2, 4, 8 and 12 weeks post treatment
Percent of responders according to the OMERACT-OARSI (Outcome Measures in Rheumatoid Arthritis Clinical Trials-Osteoarthritis Research Society International) criteria | at 4, 8 and 12 weeks post treatment
Change in patient's global assessment score | at 4, 8 and 12 weeks post treatment
Change in clinical observer's global assessment score | at 4, 8 and 12 weeks post treatment
Average weekly consumption of analgesic medications | over 12 weeks post treatment
Incidence of treatment emergent adverse events | up to 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, PhD, Study Director — Pacira Pharmaceuticals, Inc
Locations (13):
- Austria (2):
  - Graz
  - Vienna
- Canada (5):
  - Penticton, British Columbia
  - Newmarket, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Sainte-Foy, Quebec
- Spain (5):
  - Santiago de Compostela, A Coruna
  - Santander, Cantabria
  - A Coruña
  - Barcelona
  - Seville
- Southampton, United Kingdom